CLINICAL TRIAL: NCT05579067
Title: Comparative Evaluation of Functional Results and Survival Rate of Peroneus Longus Tendon - PLT and Hamstring Tendon - HT Used for Reconstruction of the Anterior Cruciate Ligament.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: eMKa MED Medical Center (Other)
Collaborators: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB-84/2022
Record Dates: First submitted 2022-03-30; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-03

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear; Knee Injuries; Knee Ligament Injury
Keywords: Injuries; Rupture; Tear; ACL; Reconstruction; Techniques
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries; Wounds and Injuries; Rupture; Lacerations

STUDY DESIGN:
Intervention Model Description: A- the use of a peroneus longus tendon autograft taken from the lower leg of the same limb and used as a graft for ACL reconstruction (anterior cruciate ligament) of the knee joint;
  B- the use of Hamstring muscle tendon autograft (Semitendonus and slender muscle) taken from the lower leg of the same limb and used as a graft for ACL reconstruction (anterior cruciate ligament) of the knee joint
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evaluation of functional results and survival rate of peroneus longus tendon used for ACLR. (Experimental)
  Interventions: Procedure: ACL Reconstruction using an autograph of the peroneus longus tendon, folded twice.
- Evaluation of functional results and survival rate of hamstring tendon used for ACL reconstruction. (Active Comparator)
  Interventions: Procedure: ACL Reconstruction using an autograph of Hamstrings muscle tendons.

INTERVENTIONS:
Procedure: ACL Reconstruction using an autograph of the peroneus longus tendon, folded twice. — The use of a peroneus longus tendon autograft taken from the lower leg of the same limb and used as a graft to reconstruct the ACL (anterior cruciate ligament) of the knee joint.
  Arms: Evaluation of functional results and survival rate of peroneus longus tendon used for ACLR.
Procedure: ACL Reconstruction using an autograph of Hamstrings muscle tendons. — The use of Hamstring muscle tendon autograft (Semitendinus and slender muscle) taken from the lower leg of the same limb and used as a graft to reconstruct the ACL (anterior cruciate ligament) of the knee joint.
  Arms: Evaluation of functional results and survival rate of hamstring tendon used for ACL reconstruction.

SUMMARY:
Comparative evaluation of functional results and survival rate of peroneus longus tendon - PLT and hamstring tendon - HT used for reconstruction of the anterior cruciate ligament.

DETAILED DESCRIPTION:
Comparison of treatment results - survival and reconstruction of autographs and functional results of the knee joint, and functional results of the ankle joint, obtained in the study groups operated using two methods:

A- the use of a long fibular tendon autograft taken from the lower leg of the same limb and used as a graft for ACL reconstruction (anterior cruciate ligament) of the knee joint; B- the use of Hamstring muscle tendon autograft (Semitendonus and slender muscle) taken from the lower leg of the same limb and used as a graft for ACL reconstruction (anterior cruciate ligament) of the knee joint.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years;
* Surgery for ACL damage to the knee joint;
* Arthroscopic surgery;
* No prior knee surgical interventions;
* No additional pathologies in this anatomical area;
* Patient informed consent to participate in research.

Exclusion Criteria:

* Age under 18 or over 65;
* Previous surgical interventions in the examined anatomical area;
* Additional pathologies in this area identified as part of preoperative diagnostics;
* Damage to the second knee joint;
* Failure to comply with the rigor of the same rehabilitation treatment protocol.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men operated on for instability of the knee joint as a result of damage to the anterior cruciate ligament.
Enrollment: 60 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-02-02 (Estimated); Study Completion 2024-02-09 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score (VAS) | 1 day
  Visual Analogue Score - subjective measure for acute and chronic pain. 100-mm VAS ratings of:
  * 0 to 4 mm can be considered no pain;
  * 5 to 44 mm, mild pain;
  * 45 to 74 mm, moderate pain;
  * 75 to 100 mm, severe pain.
Visual Analogue Score (VAS) | 3 months after procedure
  Visual Analogue Score - subjective measure for acute and chronic pain. 100-mm VAS ratings of:
  * 0 to 4 mm can be considered no pain;
  * 5 to 44 mm, mild pain;
  * 45 to 74 mm, moderate pain;
  * 75 to 100 mm, severe pain.
Visual Analogue Score (VAS) | 6 months after procedure
  Visual Analogue Score - subjective measure for acute and chronic pain. 100-mm VAS ratings of:
  * 0 to 4 mm can be considered no pain;
  * 5 to 44 mm, mild pain;
  * 45 to 74 mm, moderate pain;
  * 75 to 100 mm, severe pain.
Tegner Activity Level Scale (TAS) | 1 day
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Activity Level Scale (TAS) | 3 months after procedure
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Activity Level Scale (TAS) | 6 months after procedure
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 1 day
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 3 months after procedure
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 6 months after procedure
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
Tegner Lysholm Knee Scoring Scale | 1 day
  The Tegner Lyshom Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
  Grading the Tegner Lysholm Knee Scoring Scale:
  * <65 - poor;
  * 65-83 - fair;
  * 84-90 - good;
  * >90 - excellent.
Tegner Lysholm Knee Scoring Scale | 3 months after procedure
  The Tegner Lyshom Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
  Grading the Tegner Lysholm Knee Scoring Scale:
  * <65 - poor;
  * 65-83 - fair;
  * 84-90 - good;
  * >90 - excellent.
Tegner Lysholm Knee Scoring Scale | 6 months after procedure
  The Tegner Lyshom Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
  Grading the Tegner Lysholm Knee Scoring Scale:
  * <65 - poor;
  * 65-83 - fair;
  * 84-90 - good;
  * >90 - excellent.
Body Mass Index (BMI) | 1 day
  BMI is interpreted using standard weight status categories:
  I : below 18.5 kg/m2 - underweight;
  II : 18.5 - 24.9 kg/m2 - healthy weight;
  III : 25.0 - 29.9 kg/m2 - overweight;
  IV : 30.0 kg/m2 and above - obesity.
Body Mass Index (BMI) | 3 months after procedure
  BMI is interpreted using standard weight status categories:
  I : below 18.5 kg/m2 - underweight;
  II : 18.5 - 24.9 kg/m2 - healthy weight;
  III : 25.0 - 29.9 kg/m2 - overweight;
  IV : 30.0 kg/m2 and above - obesity.
Body Mass Index (BMI) | 6 months after procedure
  BMI is interpreted using standard weight status categories:
  I : below 18.5 kg/m2 - underweight;
  II : 18.5 - 24.9 kg/m2 - healthy weight;
  III : 25.0 - 29.9 kg/m2 - overweight;
  IV : 30.0 kg/m2 and above - obesity.
The American Orthopedic Foot and Ankle Score (AOFAS) | 1 day
  is a standardized evaluation of the clinical status of the ankle-hindfoot. It incorporates both subjective and objective information. Patients report their pain, and physicians assess alignment. The patient and physician work together to complete the functional portion.each measure is comprised of nine questions and cover three categories: Pain (40 points), function (50 points) and alignment (10 points). These are all scored together for a total of 100 points. Scores range from 0 to 100, with healthy ankles receiving 100 points.
The American Orthopedic Foot and Ankle Score (AOFAS) | 3 month after procedure
  is a standardized evaluation of the clinical status of the ankle-hindfoot. It incorporates both subjective and objective information. Patients report their pain, and physicians assess alignment. The patient and physician work together to complete the functional portion.each measure is comprised of nine questions and cover three categories: Pain (40 points), function (50 points) and alignment (10 points). These are all scored together for a total of 100 points. Scores range from 0 to 100, with healthy ankles receiving 100 points.
The American Orthopedic Foot and Ankle Score (AOFAS) | 6 month after procedure
  is a standardized evaluation of the clinical status of the ankle-hindfoot. It incorporates both subjective and objective information. Patients report their pain, and physicians assess alignment. The patient and physician work together to complete the functional portion.each measure is comprised of nine questions and cover three categories: Pain (40 points), function (50 points) and alignment (10 points). These are all scored together for a total of 100 points. Scores range from 0 to 100, with healthy ankles receiving 100 points.
Biomechanical examination | 3 months after procedure
  On the Biodex 3 System measuring device
Biomechanical examination | 6 months after procedure
  On the Biodex 3 System measuring device
Ultrasonography (USG) | 6 months after procedure
  Ultrasound examination on the apparatus with the option of elastometry
Magnetic resonance imaging (MRI) | 6 months after procedure
  1,5 Tesli

CONTACTS AND LOCATIONS:
Locations (1):
- eMKa MED Medical Center, Wroclaw, Dolnośląsk, Poland

IPD SHARING:
Plan to Share IPD: No